CLINICAL TRIAL: NCT02349451
Title: A Phase 2 Study to Investigate the Safety, Tolerability and Efficacy of ABT-122 in Subjects With Active Psoriatic Arthritis Who Have an Inadequate Response to Methotrexate
Brief Title: A Phase 2 Study to Investigate the Safety, Tolerability and Efficacy of ABT-122 in Subjects With Active Psoriatic Arthritis (PsA) Who Have an Inadequate Response to Methotrexate (MTX)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M14-197; 2014-003558-15 (EudraCT Number)
Record Dates: First submitted 2015-01-23; First posted 2015-01-28 (Estimated); Results first posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Psoriatic Arthritis
Keywords: Safety; Efficacy; Methotrexate
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Adalimumab; ABT-122

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Adalimumab (Active Comparator): Double-blind adalimumab 40 mg administered every other week (EOW) for 12 weeks
  Interventions: Biological: adalimumab
- Placebo (Placebo Comparator): Double-blind placebo administered every week (EW) for 12 weeks
  Interventions: Biological: ABT-122
- ABT-122 120 mg (Experimental): Double-blind ABT-122 120 mg administered EW for 12 weeks
  Interventions: Biological: ABT-122
- ABT-122 240 mg (Experimental): Double-blind ABT-122 240 mg administered EW for 12 weeks
  Interventions: Biological: ABT-122

INTERVENTIONS:
Biological: adalimumab
  Other Names: Humira; ABT-D2E7
  Arms: Adalimumab
Biological: ABT-122
  Other Names: remtolumab
  Arms: ABT-122 120 mg; ABT-122 240 mg; Placebo

SUMMARY:
This study is a Phase 2 randomized, double-blind, double-dummy, active- and placebo-controlled, parallel-group study designed to assess the safety, tolerability, efficacy, pharmacokinetics and immunogenicity of multiple doses of ABT-122 in participants with active PsA who are inadequately responding to MTX treatment.

ELIGIBILITY:
Inclusion Criteria:

* PsA diagnosis of at least 3 months duration prior to the date of first screening with ClASsification of Psoriatic ARthritis (CASPAR) confirmed diagnosis at Screening.
* Have active psoriasis defined by at least 1 psoriasis lesion >= 2 cm diameter in areas other than the axilla or groin.
* Have active arthritis defined by minimum disease activity criteria:

  1. >= 3 swollen joints (based on 66 joint counts) at Screening
  2. >= 3 tender joints (based on 68 joint counts) at Screening
* On a stable dose of methotrexate (MTX) defined as:

  1. Oral or parenteral treatment >= 3 months
  2. On a stable dose with an unchanged mode of application for at least 4 weeks prior to baseline
  3. Stable MTX dose of >= 10 mg/week and <= the upper limit of the applicable approved local label
  4. Can also be on stable doses of nonsteroidal anti-inflammatory drugs, sulfasalazine and/or hydroxychloroquine as long as they are also on methotrexate

Exclusion Criteria:

* Up to 30% (approximately 66 subjects) with prior exposure to a TNF inhibitor may be enrolled if the TNF inhibitor was not discontinued due to lack of efficacy or safety concerns. Subjects must be washed out for at least 5 half-lives of these drugs prior to the Baseline visit.
* Subjects on prior adalimumab may not be enrolled in the study
* Prior exposure to other non-TNF inhibitor biological disease-modifying antirheumatic drugs (DMARDs) will be permitted if the subject is washed out at least 5 half-lives of these drugs prior to the baseline visit.
* Current treatment with traditional oral/intramuscular DMARDs, including conventional synthetic DMARDs (csDMARDs; except for concomitant treatment with sulfasalazine and/or hydroxychloroquine in addition to MTX). Oral DMARDs must be washed out for at least 5 half-lives of a drug apart from MTX prior to the Baseline visit.

  a. Subject could have been exposed to prior Janus kinase (JAK) or phosphodiesterase type 4 (PDE4) inhibitors so long as they have been off therapy for at least 5 half-lives.
* Stable prescribed dose of oral prednisone or prednisone equivalent > 10 mg/day within the 30 days of the Baseline visit.
* Intra-articular or parenteral administration of corticosteroids in the preceding 4 weeks of the Baseline visit. Inhaled corticosteroids for stable medical conditions are allowed.
* Laboratory values of the following at the Screening Visit:

  1. Confirmed hemoglobin < 9 g/dL for males and < 8.5 g/dL for females
  2. Absolute neutrophil count (ANC) < 1500 mm^3, (or < 1200 cells/µL for subjects of African descent who are black)
  3. Aspartate aminotransferase or alanine aminotransferase > 1.5 x the upper limit of normal (ULN) or bilirubin >= 3 mg/dL
  4. Serum creatinine > 1.5 x the ULN
  5. Platelets < 100,000 cells/[mm^3] (10^9/L),
  6. Clinically significant abnormal screening laboratory results as evaluated by the Investigator

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2016-07-04 (Actual); Study Completion 2016-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Peloso, MD, Study Director — AbbVie

REFERENCES:
- [Derived] Khatri A, Klunder B, Peloso PM, Othman AA. Exposure-response analyses demonstrate no evidence of interleukin 17A contribution to efficacy of ABT-122 in rheumatoid or psoriatic arthritis. Rheumatology (Oxford). 2019 Feb 1;58(2):352-360. doi: 10.1093/rheumatology/key312. PMID 30376130
- [Derived] Mease PJ, Genovese MC, Weinblatt ME, Peloso PM, Chen K, Othman AA, Li Y, Mansikka HT, Khatri A, Wishart N, Liu J. Phase II Study of ABT-122, a Tumor Necrosis Factor- and Interleukin-17A-Targeted Dual Variable Domain Immunoglobulin, in Patients With Psoriatic Arthritis With an Inadequate Response to Methotrexate. Arthritis Rheumatol. 2018 Nov;70(11):1778-1789. doi: 10.1002/art.40579. PMID 29855175
- See also: Humira Prescribing info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo EW: Double-blind placebo administered every week (EW) for 12 weeks
- Adalimumab 40 mg EOW: Double-blind adalimumab 40 mg administered every other week (EOW) for 12 weeks
- ABT-122 120 mg EW: Double-blind ABT-122 120 mg administered EW for 12 weeks
- ABT-122 240 mg EW: Double-blind ABT-122 240 mg administered EW for 12 weeks
Period: Overall Study
Arm/Group | Placebo EW | Adalimumab 40 mg EOW | ABT-122 120 mg EW | ABT-122 240 mg EW
Started | 24 | 72 | 71 | 73
Completed | 24 | 71 | 69 | 72
Not Completed | 0 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: randomized participants who received at least 1 dose of study medication.
Groups:
- Placebo EW: Double-blind placebo administered EW for 12 weeks
- Adalimumab 40 mg EOW: Double-blind adalimumab 40 mg administered EOW for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo EW | Adalimumab 40 mg EOW | ABT-122 120 mg EW | ABT-122 240 mg EW | Total
Number analyzed (Participants) | 24 | 72 | 71 | 73 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (13.67) | 50.5 (12.03) | 51.0 (12.39) | 47.4 (13.77) | 49.4 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 33 | 37 | 37 | 119
  Male | 12 | 39 | 34 | 36 | 121

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology (ACR) 20 Response Rate at Week 12: ABT-122 Versus Placebo
Description: Percentage of participants with an ACR20 response, defined as at least 20% improvement (compared to baseline values) in tender and swollen joint counts and at least 20% improvement in 3 of the remaining 5 core set measures (subject global assessment of pain, subject global assessment of disease activity, physician global assessment of disease activity, subject assessment of physical function and acute phase reactant high sensitivity C-reactive protein [hsCRP]). Estimates of the 95% confidence interval of the response rates for each treatment group were calculated using the Agresti-Coull method.
Time Frame: Week 12
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug. Non-responder imputation (NRI): missing responses are imputed as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo EW | ABT-122 120 mg EW | ABT-122 240 mg EW
Number analyzed (Participants) | 24 | 71 | 73
percentage of participants | 25.0 [11.7 to 45.2] | 64.8 [53.2 to 74.9] | 75.3 [64.3 to 83.9]
Statistical Analysis 1: Comparison: Placebo EW vs ABT-122 120 mg EW; Test type: Superiority; p < 0.001, Fisher Exact — P-value is calculated by one-sided Fisher's exact test to test whether ABT-122 treatment group is superior to placebo group. The a priori statistical significance threshold is P = 0.025; response rate difference = 39.8, 95% CI 2-sided [17.2 to 57.7]
Statistical Analysis 2: Comparison: Placebo EW vs ABT-122 240 mg EW; Test type: Superiority; p < 0.001, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; response rate difference = 50.3, 95% CI 2-sided [28.1 to 67.4]

2. Secondary Outcome: ACR20 Response Rate at Week 12: ABT-122 Versus Adalimumab
Description: Percentage of participants with an ACR20 response, defined as at least 20% improvement (compared to baseline values) in tender and swollen joint counts and at least 20% improvement in 3 of the remaining 5 core set measures (subject global assessment of pain, subject global assessment of disease activity, physician global assessment of disease activity, subject assessment of physical function and acute phase reactant hsCRP). Estimates of the 95% confidence interval of the response rates for each treatment group were calculated using the Agresti-Coull method.
Time Frame: Week 12
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug. NRI: missing responses are imputed as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab 40 mg EOW | ABT-122 120 mg EW | ABT-122 240 mg EW
Number analyzed (Participants) | 72 | 71 | 73
percentage of participants | 68.1 [56.6 to 77.7] | 64.8 [53.2 to 74.9] | 75.3 [64.3 to 83.9]
Statistical Analysis 1: Comparison: Adalimumab 40 mg EOW vs ABT-122 120 mg EW; Test type: Superiority; p = 0.723, Fisher Exact — P-value is calculated by one-sided Fisher's exact test to test whether ABT-122 treatment group is superior to adalimumab group; response rate difference = -3.3, 95% CI 2-sided [-18.5 to 12.1]
Statistical Analysis 2: Comparison: Adalimumab 40 mg EOW vs ABT-122 240 mg EW; Test type: Superiority; p = 0.215, Fisher Exact — [p-value comment as in outcome 2, analysis 1]; response rate difference = 7.3, 95% CI 2-sided [-7.4 to 21.6]

3. Secondary Outcome: ACR50 Response Rate at Week 12
Description: Percentage of participants with an ACR50 response, defined as at least 50% improvement (compared to baseline values) in tender and swollen joint counts and at least 50% improvement in 3 of the remaining 5 core set measures (subject global assessment of pain, subject global assessment of disease activity, physician global assessment of disease activity, subject assessment of physical function and acute phase reactant hsCRP. Estimates of the 95% confidence interval of the response rates for each treatment group were calculated using the Agresti-Coull method.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo EW | Adalimumab 40 mg EOW | ABT-122 120 mg EW | ABT-122 240 mg EW
Number analyzed (Participants) | 24 | 72 | 71 | 73
percentage of participants | 12.5 [3.5 to 31.8] | 37.5 [27.2 to 49.1] | 36.6 [26.3 to 48.3] | 53.4 [42.1 to 64.4]
Statistical Analysis 1: Comparison: Placebo EW vs ABT-122 120 mg EW; Test type: Superiority; p = 0.021, Fisher Exact — P-value is calculated by one-sided Fisher's exact test to test whether ABT-122 treatment group is superior to placebo group; response rate difference = 24.1, 95% CI 2-sided [3.9 to 39.3]
Statistical Analysis 2: Comparison: Adalimumab 40 mg EOW vs ABT-122 120 mg EW; Test type: Superiority; p = 0.611, Fisher Exact — [p-value comment as in outcome 2, analysis 1]; response rate difference = -0.9, 95% CI 2-sided [-16.5 to 14.8]
Statistical Analysis 3: Comparison: Placebo EW vs ABT-122 240 mg EW; Test type: Superiority; p < 0.001, Fisher Exact — [p-value comment as in outcome 3, analysis 1]; response rate difference = 40.9, 95% CI 2-sided [20.1 to 55.8]
Statistical Analysis 4: Comparison: Adalimumab 40 mg EOW vs ABT-122 240 mg EW; Test type: Superiority; p = 0.039, Fisher Exact — [p-value comment as in outcome 2, analysis 1]; response rate difference = 15.9, 95% CI 2-sided [-0.3 to 31.3]

4. Secondary Outcome: ACR70 Response Rate at Week 12
Description: Percentage of participants with an ACR70 response, defined as at least 70% improvement (compared to baseline values) in tender and swollen joint counts and at least 70% improvement in 3 of the remaining 5 core set measures (subject global assessment of pain, subject global assessment of disease activity, physician global assessment of disease activity, subject assessment of physical function and acute phase reactant hsCRP. Estimates of the 95% confidence interval of the response rates for each treatment group were calculated using the Agresti-Coull method.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo EW | Adalimumab 40 mg EOW | ABT-122 120 mg EW | ABT-122 240 mg EW
Number analyzed (Participants) | 24 | 72 | 71 | 73
percentage of participants | 4.2 [0.0 to 21.9] | 15.3 [8.6 to 25.5] | 22.5 [14.3 to 33.6] | 31.5 [22.0 to 42.9]
Statistical Analysis 1: Comparison: Placebo EW vs ABT-122 120 mg EW; Test type: Superiority; p = 0.034, Fisher Exact — [p-value comment as in outcome 3, analysis 1]; response rate difference = 18.4, 95% CI 2-sided [1.5 to 29.7]
Statistical Analysis 2: Comparison: Adalimumab 40 mg EOW vs ABT-122 120 mg EW; Test type: Superiority; p = 0.185, Fisher Exact — [p-value comment as in outcome 2, analysis 1]; response rate difference = 7.3, 95% CI 2-sided [-5.8 to 19.9]
Statistical Analysis 3: Comparison: Placebo EW vs ABT-122 240 mg EW; Test type: Superiority; p = 0.004, Fisher Exact — [p-value comment as in outcome 3, analysis 1]; response rate difference = 27.3, 95% CI 2-sided [9.6 to 39.0]
Statistical Analysis 4: Comparison: Adalimumab 40 mg EOW vs ABT-122 240 mg EW; Test type: Superiority; p = 0.017, Fisher Exact — [p-value comment as in outcome 2, analysis 1]; response rate difference = 16.2, 95% CI 2-sided [2.3 to 29.3]

5. Secondary Outcome: ACRn at Week 12
Description: ACR measures percentage improvements in tender and swollen joint counts, patient assessments of pain, global disease activity and physical function, physician global assessment of disease activity and acute phase reactant. ACRn is a continuous variable based on the ACR criteria. Improvement from baseline in a component of the ACR composite variable was computed as the difference between the baseline value and the value at a given post-baseline visit. A positive value for improvement from baseline for an individual component indicates lesser severity of disease. The 95% confidence interval for mean is constructed using T-statistic with significance level alpha=5%.
Time Frame: At Week 12
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug. Last observation carried forward (LOCF): missing responses are imputed by calculation based on the last non-missing post-baseline component values.
Measure: Mean (95% Confidence Interval); unit: percentage improvement
Arm/Group | Placebo EW | Adalimumab 40 mg EOW | ABT-122 120 mg EW | ABT-122 240 mg EW
Number analyzed (Participants) | 24 | 72 | 71 | 73
percentage improvement | -20.3 [-59.6 to 19.1] | 38.2 [29.2 to 47.2] | 34.7 [25.5 to 44.0] | 48.6 [41.1 to 56.1]
Statistical Analysis 1: Comparison: Placebo EW vs ABT-122 120 mg EW; Test type: Superiority; p < 0.001, Kolmogorov-Smirnov test — Kolmogorov-Smirnov test based on the empirical distribution function is applied to get the p-value of comparing the ABT-122 treatment group with placebo group
Statistical Analysis 2: Comparison: Adalimumab 40 mg EOW vs ABT-122 120 mg EW; Test type: Superiority; p = 0.561, Kolmogorov-Smirnov test — Kolmogorov-Smirnov test based on the empirical distribution function is applied to get the p-value of comparing the ABT-122 treatment group with adalimumab group
Statistical Analysis 3: Comparison: Placebo EW vs ABT-122 240 mg EW; Test type: Superiority; p < 0.001, Kolmogorov-Smirnov test — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Adalimumab 40 mg EOW vs ABT-122 240 mg EW; Test type: Superiority; p = 0.106, Kolmogorov-Smirnov test — [p-value comment as in outcome 5, analysis 2]

6. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS28[hsCRP]) at Week 12
Description: The DAS28 (hsCRP) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, hsCRP, and general health are included in the DAS28 (hsCRP) score. Scores range from 0 to 10, with higher scores indicating more disease activity.
Time Frame: Baseline, Week 12
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug. LOCF: missing responses are imputed by calculation based on the last non-missing post-baseline component values.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo EW | Adalimumab 40 mg EOW | ABT-122 120 mg EW | ABT-122 240 mg EW
Number analyzed (Participants) | 24 | 72 | 71 | 73
units on a scale | -0.89 [-1.32 to -0.45] | -1.83 [-2.08 to -1.58] | -1.96 [-2.21 to -1.70] | -2.28 [-2.53 to -2.03]
Statistical Analysis 1: Comparison: Placebo EW vs ABT-122 120 mg EW; Test type: Superiority; p < 0.001, ANCOVA — Two-sided p-value is calculated from ANCOVA model with treatment group as the fixed factor and baseline value as the covariate; Least squares mean difference = -1.07, 95% CI 2-sided [-1.58 to -0.57]
Statistical Analysis 2: Comparison: Adalimumab 40 mg EOW vs ABT-122 120 mg EW; Test type: Superiority; p = 0.479, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least squares mean difference = -0.13, 95% CI 2-sided [-0.48 to 0.23]
Statistical Analysis 3: Comparison: Placebo EW vs ABT-122 240 mg EW; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least squares mean difference = -1.40, 95% CI 2-sided [-1.90 to -0.89]
Statistical Analysis 4: Comparison: Adalimumab 40 mg EOW vs ABT-122 240 mg EW; Test type: Superiority; p = 0.012, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least squares mean difference = -0.45, 95% CI 2-sided [-0.81 to -0.10]

7. Secondary Outcome: Change From Baseline in Psoriatic Arthritis Disease Activity Score (PASDAS) at Week 12
Description: PASDAS is a continuous compound disease activity state score determined by the combined values of tender or swollen joint counts, participant-reported outcome and hsCRP lab test. The PASDAS is unitless, with a typical score range between 0 and 10. Smaller values on PASDAS indicate a better condition; a negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo EW | Adalimumab 40 mg EOW | ABT-122 120 mg EW | ABT-122 240 mg EW
Number analyzed (Participants) | 24 | 72 | 71 | 73
units on a scale | -1.46 [-2.01 to -0.90] | -2.53 [-2.85 to -2.22] | -2.62 [-2.94 to -2.31] | -2.86 [-3.18 to -2.55]
Statistical Analysis 1: Comparison: Placebo EW vs ABT-122 120 mg EW; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least squares mean difference = -1.17, 95% CI 2-sided [-1.81 to -0.53]
Statistical Analysis 2: Comparison: Adalimumab 40 mg EOW vs ABT-122 120 mg EW; Test type: Superiority; p = 0.696, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least squares mean difference = -0.09, 95% CI 2-sided [-0.54 to 0.36]
Statistical Analysis 3: Comparison: Placebo EW vs ABT-122 240 mg EW; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least squares mean difference = -1.41, 95% CI 2-sided [-2.04 to -0.77]
Statistical Analysis 4: Comparison: Adalimumab 40 mg EOW vs ABT-122 240 mg EW; Test type: Superiority; p = 0.151, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least squares mean difference = -0.33, 95% CI 2-sided [-0.77 to 0.12]

8. Secondary Outcome: Change From Baseline in Psoriasis Target Lesion Score at Week 12
Description: Target lesion score for psoriasis in participants with psoriatic arthritis is calculated by adding the scores of plaque erythema, scaling and thickness. Scores range from 0 (no erythema or evidence of plaque thickness) to 10 (severe erythema and evidence of plaque thickness).
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo EW | Adalimumab 40 mg EOW | ABT-122 120 mg EW | ABT-122 240 mg EW
Number analyzed (Participants) | 24 | 72 | 71 | 73
units on a scale | -1.81 [-2.65 to -0.96] | -4.16 [-4.65 to -3.67] | -4.98 [-5.47 to -4.49] | -4.53 [-5.02 to -4.05]
Statistical Analysis 1: Comparison: Placebo EW vs ABT-122 120 mg EW; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least squares mean difference = -3.17, 95% CI 2-sided [-4.14 to -2.19]
Statistical Analysis 2: Comparison: Adalimumab 40 mg EOW vs ABT-122 120 mg EW; Test type: Superiority; p = 0.021, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least squares mean difference = -0.81, 95% CI 2-sided [-1.51 to -0.12]
Statistical Analysis 3: Comparison: Placebo EW vs ABT-122 240 mg EW; Test type: Superiority; p < 0.001, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least squares mean difference = -2.73, 95% CI 2-sided [-3.70 to -1.75]
Statistical Analysis 4: Comparison: Adalimumab 40 mg EOW vs ABT-122 240 mg EW; Test type: Superiority; p = 0.288, ANCOVA — [p-value comment as in outcome 6, analysis 1]; Least squares mean difference = -0.37, 95% CI 2-sided [-1.06 to 0.32]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from first dose of study drug until 70 days after the last dose of study drug (up to 21 weeks); Serious adverse events (AEs) were collected from the time informed consent was obtained (25.5 weeks).
Description: A TEAE is defined as any AE with onset or worsening reported by a participant from the time that the first dose of adalimumab or ABT-122 is administered until 5 half-lives (70 days) have elapsed following discontinuation of adalimumab or ABT-122 administration. TEAEs were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Placebo EW | Adalimumab 40 mg EOW | ABT-122 120 mg EW | ABT-122 240 mg EW
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/72 | 0/71 | 1/73
Other Adverse Events (participants affected / at risk) | 10/24 | 39/72 | 33/71 | 33/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo EW (N=24) | Adalimumab 40 mg EOW (N=72) | ABT-122 120 mg EW (N=71) | ABT-122 240 mg EW (N=73)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
SKIN ABRASION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
HEART RATE DECREASED (Investigations) | 0 | 0 | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo EW (N=24) | Adalimumab 40 mg EOW (N=72) | ABT-122 120 mg EW (N=71) | ABT-122 240 mg EW (N=73)
GRANULOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 2 | 1 | 1
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
LYMPHOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 2 | 2 | 1
PALPITATIONS (Cardiac disorders) | 0 | 1 | 0 | 0
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 1
HYDROCELE (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
BLEPHARITIS (Eye disorders) | 0 | 0 | 0 | 1
ERYTHEMA OF EYELID (Eye disorders) | 0 | 0 | 0 | 1
MYOPIA (Eye disorders) | 0 | 0 | 0 | 1
RETINAL VASCULAR DISORDER (Eye disorders) | 0 | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 1 | 1 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
FOOD POISONING (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1 | 0 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 1 | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 1 | 1
ORAL MUCOSA EROSION (Gastrointestinal disorders) | 0 | 0 | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 1
TOOTHACHE (Gastrointestinal disorders) | 0 | 1 | 1 | 1
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 1
FATIGUE (General disorders) | 0 | 2 | 1 | 1
GAIT DISTURBANCE (General disorders) | 0 | 0 | 0 | 1
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 1 | 0
INJECTION SITE BRUISING (General disorders) | 0 | 0 | 1 | 0
INJECTION SITE ERYTHEMA (General disorders) | 0 | 3 | 1 | 2
INJECTION SITE HAEMATOMA (General disorders) | 0 | 0 | 1 | 1
INJECTION SITE INDURATION (General disorders) | 0 | 0 | 0 | 1
INJECTION SITE OEDEMA (General disorders) | 0 | 1 | 0 | 1
INJECTION SITE PAPULE (General disorders) | 0 | 1 | 0 | 0
INJECTION SITE PRURITUS (General disorders) | 0 | 1 | 0 | 1
PERIPHERAL SWELLING (General disorders) | 0 | 0 | 1 | 0
VESSEL PUNCTURE SITE PHLEBITIS (General disorders) | 1 | 0 | 0 | 0
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 0 | 0 | 0 | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 0 | 0 | 1
HYPERTRANSAMINASAEMIA (Hepatobiliary disorders) | 0 | 1 | 0 | 0
ACUTE SINUSITIS (Infections and infestations) | 0 | 2 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 1 | 1 | 0
CONJUNCTIVITIS (Infections and infestations) | 0 | 0 | 0 | 1
FOLLICULITIS (Infections and infestations) | 0 | 0 | 0 | 1
FURUNCLE (Infections and infestations) | 0 | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 1 | 0 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 0 | 1 | 0
HORDEOLUM (Infections and infestations) | 0 | 0 | 1 | 0
INFLUENZA (Infections and infestations) | 0 | 3 | 0 | 1
LARYNGITIS (Infections and infestations) | 0 | 0 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 6 | 4 | 3
ORAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 1 | 1
ORAL HERPES (Infections and infestations) | 0 | 1 | 0 | 0
PARONYCHIA (Infections and infestations) | 1 | 0 | 0 | 0
PHARYNGITIS (Infections and infestations) | 0 | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 1
RHINITIS (Infections and infestations) | 1 | 0 | 0 | 1
SINUSITIS (Infections and infestations) | 1 | 0 | 1 | 1
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 | 0 | 2 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 5 | 1 | 7
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 2 | 4
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 | 0 | 1 | 0
VIRAL PHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
ANIMAL SCRATCH (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
SPLINTER (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 2 | 5 | 3
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1 | 3 | 2
BLOOD CALCIUM INCREASED (Investigations) | 0 | 0 | 1 | 0
BLOOD CHOLESTEROL INCREASED (Investigations) | 0 | 1 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 1 | 0
BLOOD PRESSURE INCREASED (Investigations) | 0 | 2 | 1 | 1
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 0 | 1 | 2 | 1
BLOOD URIC ACID INCREASED (Investigations) | 0 | 0 | 1 | 0
BODY TEMPERATURE INCREASED (Investigations) | 0 | 0 | 0 | 1
CRYSTAL URINE PRESENT (Investigations) | 0 | 0 | 1 | 1
HAEMOGLOBIN INCREASED (Investigations) | 1 | 0 | 0 | 0
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 | 2 | 0 | 1
MONOCYTE COUNT INCREASED (Investigations) | 0 | 1 | 0 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 3 | 2 | 0
TRANSAMINASES ABNORMAL (Investigations) | 0 | 0 | 0 | 1
TRANSAMINASES INCREASED (Investigations) | 0 | 0 | 2 | 0
URINE OUTPUT DECREASED (Investigations) | 0 | 0 | 1 | 0
WEIGHT INCREASED (Investigations) | 0 | 0 | 0 | 1
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 3 | 0 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 1 | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 0 | 1 | 0
SOMNOLENCE (Nervous system disorders) | 0 | 0 | 1 | 2
ANXIETY (Psychiatric disorders) | 0 | 1 | 0 | 1
DEPRESSION (Psychiatric disorders) | 0 | 1 | 0 | 0
INSOMNIA (Psychiatric disorders) | 0 | 1 | 1 | 0
STRESS (Psychiatric disorders) | 0 | 0 | 1 | 0
CRYSTALLURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0
MICTURITION URGENCY (Renal and urinary disorders) | 0 | 0 | 1 | 0
POLLAKIURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0
PROTEINURIA (Renal and urinary disorders) | 0 | 1 | 2 | 1
CATARRH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
SINUS PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
ACNE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
ECONOMIC PROBLEM (Social circumstances) | 0 | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 2 | 1 | 0
PHLEBITIS (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.